CLINICAL TRIAL: NCT03664856
Title: The Opinion of Patients With Cancer on the Claeys-Leonetti Law, on Euthanasia and the Search for Determining Factors
Brief Title: The Opinion of Patients With Cancer on the Claeys-Leonetti Law, on Euthanasia and Determining Factors
Acronym: EPAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-35
Record Dates: First submitted 2018-09-07; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Subject suffering from a locally advanced or metastatic cancer therefore falling under palliative care as defined by the definition of the French Society of Support and Palliative Care An interview will be performed
  Interventions: Other: interview

INTERVENTIONS:
Other: interview — The patient will be asked to answer the questions that the interviewer will ask him.

SUMMARY:
The law of February 2nd 2016, known as Claeys-Leonetti, reformed the legislation of the end of life. It establishes in particular a right of the patient to deep and continuous sedation, makes advance directives binding but refuses access to euthanasia. It states that artificial hydration and nutrition are treatments and not cares, which means that they can be stopped once they are deemed unnecessary, disproportionate or have no other effect than artificial maintenance of life.

While a number of personalities from all walks of life were heard during the parliamentary debate, it was found that patients were not asked about main issues under discussion. Therefore, the investigators found it useful to collect their opinions in the context of individual interviews.

A feasibility study was carried out among 40 patients, which demonstrated the feasibility of such project. This study is the subject of an article which is currently submitted to the BMC Palliative Care Journal.

The main objective is to contribute to the elaboration of the legislation on the end of life, to its adaptation to the wishes of the patients. Patients with cancer and palliative care are directly affected by the legislation on end-of-life, and it seems legitimate that these legislative provisions correspond to their expectations. The aims also to help caregivers to act in accordance with their wishes.

DETAILED DESCRIPTION:
The law of February 2nd 2016, known as Claeys-Leonetti, reformed the legislation of the end of life. It establishes in particular a right of the patient to deep and continuous sedation, makes advance directives binding but refuses access to euthanasia. It also states that artificial hydration and nutrition are treatments and not cares, which means that they can be stopped once they are deemed unnecessary, disproportionate or have no other effect than artificial maintenance of life.

While a number of personalities from all walks of life were heard during the parliamentary debate, it was found that patients were not asked about main issues under discussion. Therefore, the investigators found it useful to collect their opinions in the context of individual interviews.

A feasibility study was carried out among 40 patients, which demonstrated the feasibility of such project. This study is the subject of an article which is currently submitted to the BMC Palliative Care Journal.

The main objective is to contribute to the elaboration of the legislation on the end of life, to its adaptation to the wishes of the patients. Patients with cancer and palliative care are directly affected by the legislation on end-of-life, and it seems legitimate that these legislative provisions correspond to their expectations. The aims also to help caregivers to act in accordance with their wishes.

ELIGIBILITY:
Inclusion Criteria:

* Subject suffering from a locally advanced or metastatic cancer therefore falling under palliative care according to the definition stated by the according to the definition stated by the French Society of Support and Palliative Care
* Subject inpatient palliative care unit or identified palliative care beds or followed by a mobile palliative care team or home-based subject followed by a palliative care network or a mobile palliative care team out-of-hospital
* Subject not opposed to taking part in the study;

Exclusion Criteria:

* Subject unable to understand the purpose and conditions of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ-C15-PAL scale | 30 minutes
  The European Organization for Research and Treatment of Cancer (EORTC) questionnaire of life quality (QLQ) is a questionnaire developed to assess the quality of life of palliative (PAL) cancer care patients.
  It is a self-questionnaire, to determine the quality of life of the patient. It contains 14 items from 1 to 4. A 15th item, from 1 to 7, gives an overall score corresponding to the quality of life that the patient feels he has.
  From a minimal score (15) representing the worst quality of life until the maximal score (63) representing the best quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France

REFERENCES:
- [Derived] Evin A, Economos G, Hugues D, Gilbert E, Gracia D, Poulain P, Mateus C, Collet E, Planchet-Barraud B, Colpaert A, Perceau-Chambard E, Calvel LY, Franck C, Mallet D, Baumstarck K, Salas S. Advanced cancer patients' knowledge and opinions regarding the French law on advance directives: a multicenter cross-sectional study. Support Care Cancer. 2026 Jan 20;34(2):109. doi: 10.1007/s00520-026-10352-3. PMID 41554986
- [Derived] Salas S, Economos G, Hugues D, Gilbert E, Gracia D, Poulain P, Mateus C, Collet E, Planchet-Barraud B, Colpaert A, Perceau-Chambard E, Calvel LY, Franck C, Mallet D, Baumstarck K, Evin A. Legalisation of euthanasia and assisted suicide: advanced cancer patient opinions - cross-sectional multicentre study. BMJ Support Palliat Care. 2024 Jan 8;13(e3):e1335-e1341. doi: 10.1136/spcare-2022-004134. PMID 37536753